CLINICAL TRIAL: NCT03709160
Title: Oral dIuretics in Very Intensive Treatment, an Early Intervention in Outpatients With Heart Failure. DIVINE STUDY
Brief Title: Oral dIuretics in Very Intensive Treatment, an Early Intervention in Outpatients With Heart Failure
Acronym: DIVINE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro en Insuficiencia Cardiaca, Mexico (Other)
Responsible Party: Principal Investigator, EDUARDO CHUQUIURE-VALENZUELA MD MSc FACC, Principal Investigator, Centro en Insuficiencia Cardiaca, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-1051
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Bumetanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUMETANIDE (Experimental): we will administrated bumetanide at dosis: oral, 2mg each 8hours for seven day.
  Interventions: Drug: Bumetanide 1 MG
- INDAPAMIDE (Active Comparator): we will administrated indapamide at dosis:oral,1.5MG each 8hours for seven day.
  Interventions: Drug: Bumetanide 1 MG

INTERVENTIONS:
Drug: Bumetanide 1 MG — all patients will be taking the treatment recommended by heart failure guidelines
  Other Names: heart failure guidelines treatment

SUMMARY:
In the present study, consecutive patients, older than 18 years, of both genders will be included. The diagnosis of reduced Heart Failure (HfrEF) according to: Clinical pattern, laboratories and Cardiac imaging (ESC criteria). Treatment will be assigned in two groups: Bumetanide and another group will be received Indapamide. Each group received maximum tolerated dose for seven days with Clinical and labs evaluations will be every 48 hrs. (Face-to-face and/or telephone visits). Serum and urinary labs, EKG´s, Echo will be evaluated. Daily in-home register will made. Final points were: Mortality, Urinary failure, Clinical Impairment, Hospital admissions, Oedema. (MUCHO). All patients will be followed for 30 days.

DETAILED DESCRIPTION:
In selected patients who sign informed consent with decompensation of cardiac failure by water congestion will be allocated in two groups: Bumetanide and the other Indapamide group. Each group will be given the maximum tolerated dose for seven days with clinical evaluations every 48 hours. (Face to face and/or telephone). Clinical variables, ECG and serum and urine laboratories will be assessed finally, patients will follow up for 30 days. To identify endpoints such as: mortality, urinary failure, clinical deterioration, hospital admissions, edema. (MUCHO).

ELIGIBILITY:
Inclusion Criteria:

* 1. Older over 18 year 2. Both gender. 3. Patients are able to read, write and understand. 4.-Heart failure criteria:a) Clinical signs and symptoms b) serum NTP-proBNP: over 125pg/ml. or serum bnp: over: 35pg/ml. c) Left ventricular ejection fraction under 40% ( By any image study: echocardiogram, Tomography , MRI,Nuclear medicine.) 5. Commitment to participate in the follow-up of the present study.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with deterioration of their clinical condition that warrant rapid attention by the emergency department.
3. Patients with symptomatic hypotension by arterial pressure over; 90/50 mmHg.
4. Symptomatic heart rate disorders: tachycardia greater than 120 beats per minute or bradycardia less than 50 beats per minute.
5. Patients with respiratory impairment: by tachypnea (respiratory rate greater than 22 per min), peripheral oxygen saturation less than 90%.
6. Clinical signs or by methods of pleural effusion image that compromise the ventilatory mechanism.
7. Hormonal thyroid decontrol (thyroid hormone profile outside the reference range)
8. Serum glucose numbers greater than 140mg/DL and/or glycosylated hemoglobin greater than 6.5%.
9. Renal damage characterized by serum creatinine numbers greater than 1.5 mg/DL.
10. Alteration of the hepatic test: serum aspartate aminotransferase and/or serum alanine aminotransferase by levels greater than three times the upper limit of reference.
11. Alterations in serum electrolytes (by sodium greater 135 mmol/L or less 145 mmol; Potassium less than 3.5 mmol/L or higher 5.35 mmol/L)
12. Intolerance or allergy recognized for any diuretic.
13. Comorbidities that prevent the follow-up of treatment: (Alcoholism, drug addiction, psychiatric disorders)
14. Positive serology carriers for Hepatitis (B, C) HIV.
15. Acute myocardial infarction (with and without elevation) in the last three months.
16. History of vascular (ischemic or hemorrhagic) brain disease in the last three months.
17. Carriers of acute inflammatory and/or immunologic disease in the last three months (e.g. Active Lupus etc.)
18. Active myocarditis in the last three months
19. History of Prostatism, or recognized prostatic alterations, that impede voiding flow.
20. Terminal cancer
21. Blunt physical and cognitive deterioration that prevents optimal follow-up.
22. Cultural barriers involving limitation of communication (languages, dialects, reading and writing, etc.).
23. Not to sign informed consent

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-10-15 (Estimated)

PRIMARY OUTCOMES:
MORTALITY | 30 DAY
  HEART FAILURE DEATH, CARDIOVASCULAR DEATH, OTHER DEATH

SECONDARY OUTCOMES:
REHOSPITALIZATION | 30 DAY
  HEART FAILURE REHOSPITALIZATION, CARDIOVASCULAR REHOSPITALIZATION, OTHER REHOSPITALIZATION
URINARY FAILURE | 30 DAY
  RENAL DETERIORATION (GFR < 50%)
CLINICAL IMPAIRMENT | 30 DAY
  FUNCTIONAL CLASS DETERIORATION
OEDEMA | 30 DAY
  ABNORMAL ACCUMULATION OF FLUID (SWOLLEN ANKLE)

CONTACTS AND LOCATIONS:
Overall Officials: EDUARDO CHUQUIURE-VALENZUELA, MD MSc, Study Director — HEART FAILURE CENTER INSTITUTO NACIONAL DE CARDIOLOGIA
Locations (1):
- Centro de Insuficiencia Cardiaca Instituto Nacional de Cardiologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Individua participant data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: will be available from the publication up to 10 years after the publication
Access Criteria: Upon request addressed to principal investigator, specifying the Statistical Analysis Plan specific points you want to review

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819